CLINICAL TRIAL: NCT01227291
Title: Study With SYL040012. Tolerance and Effect on Intraocular Pressure in Subjects With IOP >= 21 mm Hg.
Brief Title: SYL040012. Tolerance and Effect on Intraocular Pressure in Subjects With Intraocular Pressure (IOP) >= 21 mm Hg
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYL040012_II
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; IOP; siRNAs; RNAi; beta inhibitor
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SYL040012 (Experimental): SYL040012 Ophthalmic drop administration
  Interventions: Drug: SYL040012

INTERVENTIONS:
Drug: SYL040012 — SYL040012 ophthalmic drops, daily single dose administration
  Other Names: No additional names

SUMMARY:
The aim of this study is to evaluate the tolerance and effect on unmedicated subjects with elevated IOP.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the tolerance and effect on unmedicated subjects with elevated IOP. An unmedicated subject is considered a person without any IOP/glaucoma treatment at least one month before recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* >/= 18 years of age with elevated IOP with OAG diagnosis.
* Subjects must provide signed informed consent prior to participation in any study-related procedures
* IOP >/= 21 mmHg and < 30 mmHg in three different assessment days.
* Normal Ocular test (in both eyes):

  * Visual field: 24-2 or equivalent
  * Normal OCT
  * BCVA: >/= 0,5 (20/40) Snellen scale, or </=0.3 LogMar.
  * Normal Schirmer Test .
  * Normal funduscopy.

Exclusion Criteria:

* Pregnant or breastfeeding females or those with a positive pregnancy test. Females of childbearing potential who will not use a medically acceptable contraceptive method from selection and during the hole study.
* Current relevant disease, including respiratory disease, cardiovascular, endocrine, neurological, hematological, renal, neoplastic, hepatopathy, gastrointestinal distress, hypertension or infectious acute processes.
* Previous chronic processes or with rebound characteristics that could interfere with the study according to the investigator's judgment.
* Having used betablockers and corticoids sporadically in the last 15 days whichever the route of administration.
* Previous eye refractive surgery
* Subjects with visual alteration with more than 3 dioptres for hypermetropy and/or astigmatism.
* Use of contact lenses during the last 7 days before starting the treatment.
* Subjects who has participated in a clinical trial during the past 2 months before study entry.
* Analytic alterations medically relevant, at investigator judgment.
* Positive results in test drug abuse during selection period.
* Subjects with at least 2 visual fields or fiber layer measured in two different days abnormals
* History of ocular infection or inflammation within the past 3 months
* Pachymetry(in the middle of the cornea) >600 microm or < 500 microm.
* Subjects with IOP associated to close angle glaucoma
* History of chronic or severe acute ocular disease (i.e. scleritis, uveitis, blepharitis, conjunctivitis or herpes simplex virus)
* History of intolerance to any of the components of the drug formulation
* Subjects with previous iridotomy with IOP related with close angle glaucoma.
* Previous ocular surgery in glaucoma
* Corneal refractive surgery (e.g., keratotomy, PRK, LASIK, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Tolerance on ocular surface (ocular and conjunctiva) | 7 days + 24 hours
  Local Tolerance and ocular surface(cornea and conjunctival) on the area of administration 24 hours after last administration of multiple dose during 7 days of administration. It will be performed using a slit lamp which will be performed before, during and after the administration at established times. Adverse events will be registered and the determination of subjective tolerance will use the visual analogical scale (VAS) in cases where a subjects refers them.

SECONDARY OUTCOMES:
Tolerance, Adverse events, Pharmacokinetics and effect | 11 days
  Local Tolerance on the area of administration at 1 hour and 96 hours after the last administered dose: corneal pachymetry, rest of anterior exploration of the eye, visual acuity, eye fundus, clinical exam (including physical exploration, vital signs, analytical blood and urine test, and ECG.
  Other parameters: analytics, VAS evaluation, Evaluation of adverse event appearance Pharmacokinetics: SYL040012 blood absorption will be evaluated after topical ocular administration Effect on IOP

CONTACTS AND LOCATIONS:
Overall Officials: Javier Moreno, MD, PhD, Principal Investigator — Clinica Universidad de Navarra; Francisco Muñoz, MD, PhD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (2):
- Spain (2):
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Clinica Universidad Navarra, Pamplona, Navarre